CLINICAL TRIAL: NCT03788473
Title: "Periodontal Disease as a Possible Risk Factor for Complications During Pregnancy and Childbirth
Acronym: PERIOEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Doctor of science in Nursing, Universidad de Granada
Other Study IDs: BECOME
Record Dates: First submitted 2018-12-06; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Periodontitis During Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control.: Healthy Pregnant
- Case.: Pregnant with Periodontal Disease

SUMMARY:
Pregnancy is a physiological state that is part of the reproductive life of women, establishing their fertile age between 15 and 45 years mainly. This stage will not only mark the birth of the baby but also cause various changes both immunological and physiological, to accommodate the growing fetus.

Maternal periodontitis has direct and indirect potential to influence the health of the fetus-maternal unit. According to the literature reviewed, the first evidence that oral bacteria influenced pregnancy outcomes was reported by Collins et al. The injection of P. gingivalis into pregnant hamsters caused intrauterine growth retardation and smaller fetuses, together with an increase in the levels of proinflammatory mediators (IL-1b and PGE2) in the amniotic fluid.

Two hypotheses have been pointed out regarding the link between oral health and the adverse outcome of pregnancy. The first states that periodontal disease causes abnormal systemic immune changes, leading to complications in pregnancy. While the second hypothesis suggests that oral bacteria directly colonize the placenta, causing localized inflammatory responses, resulting in prematurity and other adverse outcomes.

DETAILED DESCRIPTION:
Pregnancy is a physiological state that is part of the reproductive life of women, establishing their fertile age between 15 and 45 years mainly. This stage will not only mark the birth of the baby but also cause various changes both immunological and physiological, to accommodate the growing fetus. In Spain, according to the Spanish National Institute of Statistics (INE), a total of 195,555 births were registered in 2017.

However the arrival of the birth sometimes has adverse results for the mother and baby, such as low birth weight (<2500 g), premature birth (<37 weeks), growth restriction (weight for gestational age), preeclampsia, spontaneous abortion and / or inanimate birth. Some of these results occur together, and it is not clear if they share common mechanisms.

According to the WHO, every year around 15 million babies are born in the world before they reach term, that is, more than 1 in 10 births. Of them approximately, one million premature children die every year due to complications in childbirth. As well as every day about 830 women die from complications related to pregnancy or childbirth. While 75% of maternal deaths are due, among other causes, to gestational hypertension (preeclampsia and eclampsia).

The most common risk factor associated with premature birth is the previous history of premature birth. Other less prevalent factors are the short interval between pregnancies, assisted reproduction procedures, multiple gestation and infectious diseases such as periodontitis.

Maternal periodontitis has direct and indirect potential to influence the health of the fetus-maternal unit. According to the literature reviewed, the first evidence that oral bacteria influenced pregnancy outcomes was reported by Collins et al. The injection of P. gingivalis into pregnant hamsters caused intrauterine growth retardation and smaller fetuses, together with an increase in the levels of proinflammatory mediators (IL-1b and PGE2) in the amniotic fluid.

In humans, the first clinical study of the association between adverse pregnancy outcomes and periodontal status was a case-control study by Offenbacher et al. These authors concluded that the woman with periodontitis presented an almost 8 times greater risk of presenting a preterm delivery / low birth weight of the newborn than the periodontally healthy woman.

Two hypotheses have been pointed out regarding the link between oral health and the adverse outcome of pregnancy. The first states that periodontal disease causes abnormal systemic immune changes, leading to complications in pregnancy. While the second hypothesis suggests that oral bacteria directly colonize the placenta, causing localized inflammatory responses, resulting in prematurity and other adverse outcomes.

In 2013 it was reported that low birth weight, premature birth and preeclampsia were associated with maternal periodontitis. However, this association was moderate in relation to other studies, probably due to differences in the study population, the different means of periodontal evaluation used and the classification of periodontal disease that was used. The authors of this study, argued that the association of periodontitis and adverse pregnancy outcomes are explained by two main routes, a direct one, in which the oral microorganisms and / or their components reach the fetoplacental unit and another indirect, in the that inflammatory mediators circulate and impact the fetal-placental unit.

Therefore, according to the direct route, oral microbiota during pregnancy plays an important role in adverse obstetric outcomes. A recent meta-analysis of 22 studies that included 12047 pregnant women showed, by partially analyzing the oral microbiota, that women with periodontitis had an increased risk of preterm birth and of giving birth to a low birth weight baby.

The indirect route has also been studied by other authors, who reported that there was a positive association between inflammatory mediator levels of gingival crevicular fluid and adverse outcomes of pregnancy / preterm birth, but the results should be interpreted with caution due to heterogeneity and variability between studies However, some authors have not shown differences in the anaerobic bacterial profile or commensals among mothers with periodontitis, despite the fact that they observe local placental factors, such as the nature of the inflammatory infiltrate and the slightly higher expression of COX2 in women with these results. Adverse effects of pregnancy are related to a subclinical proinflammatory state that could contribute to triggering premature birth. In this regard Penova et al. they did not observe changes in the results related to pregnancy, although the severity of the periodontal disease was significantly associated with an increased risk of babies born small for gestational age. They highlighted that the treatment of PE in pregnancy reduces the levels of some inflammatory mediators in the gingival crevicular fluid, improving dental parameters but without obvious effects on the outcome of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 12 weeks.
* Pregnant women who consent to participate in the study by signing informed consent.

Exclusion Criteria:

* Pregnant with less than 6 teeth.
* Pregnant women who have been treated for Periodontal Disease in the last 6 months. -E Multiple branches.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Our research project "PERIOEM Study", is part of the BECOME framework project (Behavior of biomarkers (lipid profile and prolactin) during pregnancy and lactation through a biological multiparadigm model), whose main objective is to determine the evolution of the lipid profiles during pregnancy, to create a biological predictive model, which establishes thresholds above which, the increase of biomarkers constitutes a risk marker related to the development of diseases during pregnancy, childbirth and lactation. The BECOME study is registered in Clinical Trial NCT02811172; which obtained the suitability by the ethics committee on April 28, 2015.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-07-26 (Estimated); Study Completion 2021-11-26 (Estimated)

PRIMARY OUTCOMES:
CAOD | 9 months
  CAOD Index: 0: Absent or Great Destruction 1: Caries 2: Closed. It will be calculated: C + A + O.
Bleeding on probing | 9 months
  Ainamo and Bay index modified for bleeding on probing: when inserting the probe into the groove if: 0- does not bleed; 1-bleed It will be computed according to the following formula: number of bleeding points between the number of points examined per 100.
Presence of plate | 9 months
  Index of Silness and Löe: If when passing the probe: 0, there is no plate; 1, plate when passing the probe; 2, plate with the naked eye; 3, abundant plaque around the tooth even with tartar. It will be calculated by adding the values obtained for each tooth, among the number of teeth present.
Periodontal insertion level | 9 months
  Distance of the cementoenamel line to the bottom of the periodontal pocket (probing depth + recession, or probing depth - hyperplasia). It will be measured in 6 sites per tooth (mesial-vestibular, vestibular, disto-vestibular and palatal / lingual-distal, palatal / lingual, palatal / lingual-mesial).
Depth of stock | 9 months
  Distance from the gingival margin to the bottom of the periodontal pocket (junctional epithelium). It will be measured with a millimetric probe. It will be measured in 6 sites per tooth (mesial-vestibular, vestibular, disto-vestibular and palatal / lingual-distal, palatal / lingual, palatal / lingual-mesial).
Periodontal disease | 9 months
  Periodontitis was diagnosed when the loss of buccal epithelial attachment (vestibular-palatal) was greater than 3 mm and depth of the pouch greater than or equal to 3 mm in 2 teeth or more.

CONTACTS AND LOCATIONS:
Overall Officials: María José Aguilar Cordero, Profesora, Study Director — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain